CLINICAL TRIAL: NCT03071601
Title: Prospective Evaluation of Topical Analgesia Using a Lidocaine/Prilocaine Cream for Laceration Repair in the Emergency Department
Brief Title: Prospective Evaluation of Topical Analgesia for Laceration Repair in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHM-2016-S2/04
Record Dates: First submitted 2017-02-17; First posted 2017-03-07 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Pain, Acute; Laceration
Keywords: Laceration; Suture; Topical anesthesia; Lidocaine
MeSH Terms: conditions — Acute Pain; Lacerations | interventions — Lidocaine; Epinephrine; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical anesthesia (Experimental): Topical anesthesia using a cream containing 2.5% Lidocaine and 2.5% Prilocaine applied for at least 30 minutes before laceration repair.
  Interventions: Drug: Lidocaine-Prilocaine Cream 2.5-2.5%
- Subcutaneous injection anesthesia (Experimental): Local anesthesia by a subcutaneous injection of a solution containing 1% Lidocaine and 0.005 mg/mL Epinephrine in the minutes before laceration repair.
  Interventions: Drug: Lidocaine 1% Epinephrine 0.005mg/mL solution

INTERVENTIONS:
Drug: Lidocaine-Prilocaine Cream 2.5-2.5% — Topical anesthesia using a cream containing 2.5% Lidocaine and 2.5 % Prilocaine for at least 30 minutes on and around the wound before suture
  Arms: Topical anesthesia
Drug: Lidocaine 1% Epinephrine 0.005mg/mL solution — Local anesthesia by subcutaneous injection of a solution containing 1% Lidocaine and 0.005mg/mL Epinephrine in and around the wound in the minutes preceding the suture of the wound
  Arms: Subcutaneous injection anesthesia

SUMMARY:
The purpose of this study is to determine if topical analgesia using a lidocaine and prilocaine cream improves pain scores compared to the usual local anesthesia using subcutaneous 1% lidocaine and adrenalin injected near the laceration.

DETAILED DESCRIPTION:
A prospective randomized open clinical trial conducted in two high volume emergency departments in France.

Adult patients presenting for laceration repair by suture will be allocated, after consent is obtained, on a one to one basis using a randomisation by minimisation method.

126 patients are expected to enrol in the study.

ELIGIBILITY:
Inclusion Criteria:

* Superficial skin laceration requiring a suture

Exclusion Criteria:

* Known allergy to lidocaine
* Mucous membrane or eye wound
* Nose, ear or perineal wound
* Active hemorrhage in the wound
* Dirty or infected wound
* Wound requiring operation room management
* Distracting pain in an other location
* Intoxicated or comatose patient
* Patient Under guardianship
* Contra-indication to Lidocaine/Prilocaine cream: hypersensitivity, glucose-6-phosphate deficiency, idiopathic methemoglobinemia
* Neurologic disorder affecting pain sensitivity
* Dementia
* Pregnancy, breast feeding, absence of contraceptive measures for women of childbearing age
* Absence of signed informed consent
* Inclusion in an other interventional clinical protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum pain | 60 minutes
  Maximum pain on the numerical pain scale (0-10) during laceration management (anesthesia, exploration and suture of the laceration).

SECONDARY OUTCOMES:
Patient satisfaction | 60 minutes
  Patient satisfaction relating to the pain management measured on a four point Likert scale.
Topical anesthesia failure rate | 60 minutes
  Percentage of patients in the intervention group who required additional anesthesia by subcutaneous injection of Lidocaine/Epinephrine
Pain management during the various stages of care | 60 minutes
  Maximum pain measured on the numerical pain scale (0-10) measured on admission to the emergency department, during the wait for laceration treatment, during the wound cleansing for the intervention group and during anesthesia for the control group, during suture.
Management duration | 60 minutes
  Mean duration of management between admission to the emergency department and discharge.
Adverse effects | 15 days
  Evaluation of adverse effects due to the anesthesia technique (e.g. allergic reactions) by a telephone interview 15 days after initial management
Wound healing | 15 days
  Evaluation of the quality of wound healing during a telephone interview by identifying signs of wound infection and/or wound reopening.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Fonsegrive, MD, Principal Investigator — Centre Hospitalier le Mans
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire Angers, Angers
  - Centre Hospitalier Le Mans, Le Mans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McNulty RJ, Handley TP, Devlin MF. Reducing the need for general anaesthesia in children: use of LAT gel in treating facial lacerations. Br J Oral Maxillofac Surg. 2013 Sep;51(6):e130-1. doi: 10.1016/j.bjoms.2012.04.259. Epub 2012 Jun 12. PMID 22694845
- [Result] White NJ, Kim MK, Brousseau DC, Bergholte J, Hennes H. The anesthetic effectiveness of lidocaine-adrenaline-tetracaine gel on finger lacerations. Pediatr Emerg Care. 2004 Dec;20(12):812-5. doi: 10.1097/01.pec.0000148029.61222.9f. PMID 15572968